CLINICAL TRIAL: NCT04058938
Title: A Randomized Control Trial of Patient Education on Pain Control in Breast Surgery
Brief Title: Pain in Breast Surgery Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Katie Egan, Plastic Surgery Resident, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 00141330
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Opioid Use; Pain, Postoperative
Keywords: opioid use; breast reconstruction; pain control; mastectomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: All study participants received a study folder with information about the study and consent; the instrument was included in this folder for the intervention group. The control group received standard of care, including standard patient counseling from the surgical teams. In conjunction with oncologic psychology and plastic surgery, an instrument was developed to be provided as a single-paged paper handout to the intervention group. The instrument included information about expectations for pain control, information about the pain scale, and examples of opioid and adjunct medications which may be used as part of a multi-modal approach to pain control during the perioperative period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study participants were not informed of randomization, and providers involved in patient care, consent, and postoperative questionnaire administration were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The control group received standard of care, including standard patient counseling from the surgical teams.
  Interventions: Behavioral: Control
- Intervention (Experimental): In conjunction with oncologic psychology and plastic surgery, an instrument was developed to be provided as a single-paged paper handout to the intervention group. The instrument included information about expectations for pain control, information about the pain scale, and examples of opioid and adjunct medications which may be used as part of a multi-modal approach to pain control during the perioperative period.
  Interventions: Behavioral: Educational handout instrument

INTERVENTIONS:
Behavioral: Educational handout instrument — The handout was single-paged (front and back), and was titled Pain After Surgery: What to Expect. The handout starts with information on rating pain and expectations for control of pain, not complete absence of pain, after surgery. Mutli-modal approach to pain control is then discussed, including pharmacologic and non-pharmacologic methods that may be used for pain control by the perioperative team and postoperatively.
  Arms: Intervention
Behavioral: Control — Standard patient counseling
  Arms: Control

SUMMARY:
This study will be a randomized control trial providing an educational component to study participants and a pre-operative and post-operative survey with a goal to show an improvement in pain control, decrease in narcotic use, and increase in patient knowledge in the study group.

DETAILED DESCRIPTION:
The use of opioid pain medications in surgical patients is contributing to an epidemic of opioid pain medication use. It is known that the quality of pain control after surgery is a large factor of the patient's perception of their experience. However, little research has been done to improve pain control in plastic surgery patients. To the investigators knowledge, no study has yet looked at education of breast surgery patients to improve pain experience. The study goal is to survey breast surgery patients in the Plastic Surgery department before and after surgery to evaluate the participants experience with pain and pain medications. Half of the participants in the study will be randomized to receive an information sheet about pain control at the participants pre-operative appointment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients presenting for the first stage of breast reconstruction using tissue expanders
* Patients 18 years of age and older

Exclusion Criteria:

* Male patients
* Patients under age 18
* Patients who have had previous breast reconstruction or tissue expansion
* Patients who are not able to read English will be excluded from this study as the study materials will be in written English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be female patients undergoing mastectomy and breast reconstruction to be eligible for the study.
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 1-2 weeks
  Opioid consumption will be calculated from patient report of remaining narcotics at the postoperative appointment and the total opioid amount prescribed, from the medical record.

SECONDARY OUTCOMES:
Pain control: survey | 1-2 weeks
  Patient report of subjective and objective pain control after surgery will be collected on a postoperative survey. Objective pain control will be scored by asking patients to circle a pain score on a scale of 0 to 10. This is a continuous scale used to score pain with 0 being no pain and 10 being the worst pain. Subjective pain will be rated by asking participants to state yes or no for control of pain and state yes or no if pain interfered with walking, sleeping, and activities of daily living.

OTHER OUTCOMES:
Patient knowledge of pain control | 1-2 weeks.
  Patient reported knowledge of pain control will be collected on the preoperative and postoperative survey. Patients will be asked to circle yes or no to feeling like the participant had enough information about pain control and about surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Korentager, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No